CLINICAL TRIAL: NCT04099316
Title: Effects of Eccentric-based Training on Muscle Strength and Physical Function in Older Adults
Brief Title: Effects of Eccentric Training Intervention in Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Principal Investigator, Jae-Young Lim, Professor, Department of Rehabilitation Medicine, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: B-1705-397-004
Record Dates: First submitted 2019-05-16; First posted 2019-09-23 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Sarcopenia
Keywords: Aging; Eccentric training; Muscle strength; Physical function; Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Older adults (Experimental): Older adults (Over the 60 years), Subjects did not suffer from musculoskeletal or metabolic diseases.
  Interventions: Device: Eccentric exercise
- Older adults-Control (Experimental): Older adults (Over the 60 years), Subjects did not suffer from musculoskeletal or metabolic diseases.
  Interventions: Device: Conventional resistance exercise
- No intervention (No Intervention): Metabolic diseases, Hypertension (150/90mmHg), Myocardial infarction within 6 months. Fractures within 6 months.

INTERVENTIONS:
Device: Eccentric exercise — Eccentric exercise with Eccentron electronic device. Exercise intervention: The exercise intervention is performed to twice a week (Total 8 weeks). Exercise intensity is gradually increased to the number of times by divided into two stages (1-4 weeks; 1st stage),(5-8 weeks; 2nd stage).
  Arms: Older adults
Device: Conventional resistance exercise — Leg press exercise with leg press machine. Exercise intervention: The exercise intervention is performed to twice a week (total 8 weeks). Exercise intensity is gradually increased to the number of times by divided into two stages (1-4 weeks; 1st stage), (5-8 weeks; 2nd stage).
  Arms: Older adults-Control

SUMMARY:
Sarcopenia leads to loss of muscle mass and muscle strength during the aging process. It has been reported that eccentric training has some positive effects on the preservation of eccentric strength, with less delayed onset muscle soreness (DOMS) in older groups, and lower metabolic costs.

DETAILED DESCRIPTION:
This is prospective study. The goals of this study are to:

1. Examine the effects of eccentric training on physical function (gait speed, stair climb, chair stand) in older adults.
2. Examine the effects of eccentric training on muscle strength (Isometric strength, Isokinetic strength, power) in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who can agree voluntarily
* Older men/women: Age (60 - 80 yrs)

Exclusion Criteria:

* Uncontrolled hypertension
* Acute coronary syndrome
* Subjects who took drugs which can affects neuromuscular system
* Subjects who cannot agree voluntarily

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2017-07-20 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-10-31 (Estimated)

PRIMARY OUTCOMES:
Gait speed | Change from baseline gaitspeed at 8 weeks
  An examiner used a stopwatch to time how long it took subjects to walk along a marked tape. The Kinect device was used to measure gait speed.
Stair climb | Change from baseline stair climb at 8 weeks
  Subjects were measured on eight 17-cm stairs twice, requiring a step by step pattern, where the timer activated when the first contact was made at the first step and ended when the contact occurred at the last step before and after the 8 weeks of exercise training.
Chair stand | Change from baseline chair stand at 8 weeks
  Subjects had to get up from a chair measuring 41 cm in height with a flat seat. Subjects were asked to stand up and sit down 5 times as quickly as possible with their arms folded across the chest. They stood up until full extension was observed at the trunk and lower limb joints, and returned to a seated position with their back fully supported at the back of the chair.

SECONDARY OUTCOMES:
Isokinetic knee strength | Change from baseline isokinetic knee strength at 8 weeks
  The isokinetic was measured using a baltimore therapeutic equipment (BTE) Primus RS (BTE Tech., Hanover, MD, USA). The subject performed a 60 degree per second knee flexion and extension five times. Each isokinetic contraction was performed through a full range of motion.Before each subject began the isokinetic test, the subject warmed up using a 50-60% knee extension/flexion once.
  Isokinetic knee strength is measured in as peak torque achieved on an isokinetic dynamometer (BTE PrimusRS, BTE tech, MD, USA) at 60 degree per second.
Isometric knee strength | Change from baseline isometric knee strength at 8 weeks
  Isometric knee strength was measured using a baltimore therapeutic equipment (BTE) Primus RS (BTE Tech., Hanover, MD, USA). The subject was asked to sit on the treatment chair and a standard stabilization strap was placed on the upper ankle. The knee was kept at 90 degree flexion, and the foot was positioned in dorsi flexion. The subject's hands were placed on the edge of the side of the chair and the trunk, hips, and mid-thigh were stabilized in the chair by the straps.
Power | Change from baseline power at 8 weeks
  The test used same machine as the isometric and isokinetic tests. The ankle was placed in a neutral position, and the subjects performed a range of motion for 10 seconds, once. After the warm up, knee extension and flexion were performed as quickly as possible during a period of 10 seconds.
  Isokinetic knee strength is measured in as peak torque achieved on an isokinetic dynamometer (BTE PrimusRS, BTE tech, MD, USA) at 60 degree per second.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, Geyonggi, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roig M, Macintyre DL, Eng JJ, Narici MV, Maganaris CN, Reid WD. Preservation of eccentric strength in older adults: Evidence, mechanisms and implications for training and rehabilitation. Exp Gerontol. 2010 Jun;45(6):400-9. doi: 10.1016/j.exger.2010.03.008. Epub 2010 Mar 18. PMID 20303404
- [Background] Frontera WR, Hughes VA, Krivickas LS, Roubenoff R. Contractile properties of aging skeletal muscle. Int J Sport Nutr Exerc Metab. 2001 Dec;11 Suppl:S16-20. doi: 10.1123/ijsnem.11.s1.s16. No abstract available. PMID 11915915
- [Background] Frontera WR, Reid KF, Phillips EM, Krivickas LS, Hughes VA, Roubenoff R, Fielding RA. Muscle fiber size and function in elderly humans: a longitudinal study. J Appl Physiol (1985). 2008 Aug;105(2):637-42. doi: 10.1152/japplphysiol.90332.2008. Epub 2008 Jun 12. PMID 18556434
- [Background] Cadore EL, Rodriguez-Manas L, Sinclair A, Izquierdo M. Effects of different exercise interventions on risk of falls, gait ability, and balance in physically frail older adults: a systematic review. Rejuvenation Res. 2013 Apr;16(2):105-14. doi: 10.1089/rej.2012.1397. PMID 23327448
- [Background] Chen TC, Tseng WC, Huang GL, Chen HL, Tseng KW, Nosaka K. Superior Effects of Eccentric to Concentric Knee Extensor Resistance Training on Physical Fitness, Insulin Sensitivity and Lipid Profiles of Elderly Men. Front Physiol. 2017 Apr 10;8:209. doi: 10.3389/fphys.2017.00209. eCollection 2017. PMID 28443029
- [Background] Dias CP, Toscan R, de Camargo M, Pereira EP, Griebler N, Baroni BM, Tiggemann CL. Effects of eccentric-focused and conventional resistance training on strength and functional capacity of older adults. Age (Dordr). 2015 Oct;37(5):99. doi: 10.1007/s11357-015-9838-1. Epub 2015 Sep 15. PMID 26374635
- [Background] Enoka RM. Eccentric contractions require unique activation strategies by the nervous system. J Appl Physiol (1985). 1996 Dec;81(6):2339-46. doi: 10.1152/jappl.1996.81.6.2339. PMID 9018476
- [Background] Gault ML, Willems ME. Aging, functional capacity and eccentric exercise training. Aging Dis. 2013 Sep 25;4(6):351-63. doi: 10.14336/AD.2013.0400351. PMID 24307968
- [Background] Hanson ED, Srivatsan SR, Agrawal S, Menon KS, Delmonico MJ, Wang MQ, Hurley BF. Effects of strength training on physical function: influence of power, strength, and body composition. J Strength Cond Res. 2009 Dec;23(9):2627-37. doi: 10.1519/JSC.0b013e3181b2297b. PMID 19910811
- [Background] LaStayo P, Marcus R, Dibble L, Wong B, Pepper G. Eccentric versus traditional resistance exercise for older adult fallers in the community: a randomized trial within a multi-component fall reduction program. BMC Geriatr. 2017 Jul 17;17(1):149. doi: 10.1186/s12877-017-0539-8. PMID 28716003
- [Background] Lim JY. Therapeutic potential of eccentric exercises for age-related muscle atrophy. Integr Med Res. 2016 Sep;5(3):176-181. doi: 10.1016/j.imr.2016.06.003. Epub 2016 Jun 18. PMID 28462115
- [Background] Mueller M, Breil FA, Vogt M, Steiner R, Lippuner K, Popp A, Klossner S, Hoppeler H, Dapp C. Different response to eccentric and concentric training in older men and women. Eur J Appl Physiol. 2009 Sep;107(2):145-53. doi: 10.1007/s00421-009-1108-4. Epub 2009 Jun 20. PMID 19543908
- [Background] Orer GE, Guzel NA, Arslan E. Recovery levels after eccentric and concentric loading in maximal force. J Phys Ther Sci. 2016 Jun;28(6):1743-7. doi: 10.1589/jpts.28.1743. Epub 2016 Jun 28. PMID 27390407
- [Background] Raj IS, Bird SR, Westfold BA, Shield AJ. Effects of eccentrically biased versus conventional weight training in older adults. Med Sci Sports Exerc. 2012 Jun;44(6):1167-76. doi: 10.1249/MSS.0b013e3182442ecd. PMID 22143107
- [Background] Roig M, O'Brien K, Kirk G, Murray R, McKinnon P, Shadgan B, Reid WD. The effects of eccentric versus concentric resistance training on muscle strength and mass in healthy adults: a systematic review with meta-analysis. Br J Sports Med. 2009 Aug;43(8):556-68. doi: 10.1136/bjsm.2008.051417. Epub 2008 Nov 3. PMID 18981046
- [Background] Symons TB, Vandervoort AA, Rice CL, Overend TJ, Marsh GD. Effects of maximal isometric and isokinetic resistance training on strength and functional mobility in older adults. J Gerontol A Biol Sci Med Sci. 2005 Jun;60(6):777-81. doi: 10.1093/gerona/60.6.777. PMID 15983182
- [Background] Vaczi M, Nagy SA, Koszegi T, Ambrus M, Bogner P, Perlaki G, Orsi G, Toth K, Hortobagyi T. Mechanical, hormonal, and hypertrophic adaptations to 10 weeks of eccentric and stretch-shortening cycle exercise training in old males. Exp Gerontol. 2014 Oct;58:69-77. doi: 10.1016/j.exger.2014.07.013. Epub 2014 Jul 23. PMID 25064038